CLINICAL TRIAL: NCT01465672
Title: Copeptin as a Diagnostic Marker in the Management of Neurosurgical Patients With Disturbance of Water Homeostasis
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Kantonsspital Aarau (Other)
Responsible Party: Principal Investigator, Mirjam Christ-Crain, Leitende Aerztin, Prof. Dr. med., University Hospital, Basel, Switzerland
Other Study IDs: COOP Study
Record Dates: First submitted 2011-10-28; First posted 2011-11-07 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Pituitary Adenoma
Keywords: copeptin; SIADH; Diabetes insipidus; transphenoidal pituitary adenoma resection; pituitary adenoma; tumors close to pituitary gland; tumors close to hypothalamus
MeSH Terms: conditions — Pituitary Neoplasms; Diabetes Insipidus; Inappropriate ADH Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- neurosurgical patients: Patients undergoing transphenoidal pituitary adenoma resection and patients with transcranial surgery of tumors close to the pituitary gland and hypothalamus.

SUMMARY:
Water imbalance and consecutive electrolyte disturbances are common in the postoperative course of neurosurgical patients after pituitary surgery. Diabetes insipidus (DI) may complicate the postoperative course in as many as 30% of patients. Early and accurate diagnosis of water and electrolyte disturbances postoperatively is important for an adequate fluid and drug administration. However, identifying the causes is challenging/ ambiguous in clinical practice. Levels of antidiuretic hormone (ADH) might contribute to a straightforward diagnosis, though, its measurement is cumbersome. ADH is derived from a larger precursor peptide along with copeptin, which is a more stable peptide directly mirroring the production of ADH. Copeptin can be assayed readily in plasma. Aim: To investigate whether copeptin can accurately diagnose postoperative disturbances of water homeostasis (i.e. Diabetes insipidus and SIADH) in a cohort of patients undergoing intracranial tumor surgery.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who undergo surgery for an intra- or suprasellar lesion, either by craniotomy or by transphenoidal resection.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing transphenoidal pituitary adenoma resection and patients with transcranial surgery of tumors close to the pituitary gland and hypothalamus.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2011-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy, i.e. difference of copeptin levels between patients without and patients with postoperative DI, of copeptin in the diagnosis of water disturbance in neurosurgical patients | daily during hospital stay of the patient, on average 1 week
  daily blood sampling will allow to diagnose DI or SIADH during hospital stay. Copeptin levels will be compared between patients with uncomplicated postoperative course and patients with development of DI or SIADH.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - University Hospital Basel, Basel, Basel
  - Kantonsspital Aarau, Aarau

REFERENCES:
- [Derived] Winzeler B, Zweifel C, Nigro N, Arici B, Bally M, Schuetz P, Blum CA, Kelly C, Berkmann S, Huber A, Gentili F, Zadeh G, Landolt H, Mariani L, Muller B, Christ-Crain M. Postoperative Copeptin Concentration Predicts Diabetes Insipidus After Pituitary Surgery. J Clin Endocrinol Metab. 2015 Jun;100(6):2275-82. doi: 10.1210/jc.2014-4527. Epub 2015 Apr 29. PMID 25923040